CLINICAL TRIAL: NCT06967402
Title: Comparative Clinical Efficacy and Microbiological Effects of Two Oral Antiseptics Used as an Adjuvant in the Treatment of Severe Periodontitis
Brief Title: Comparative Effects of Two Oral Antiseptics Used as an Adjuvant in the Treatment of Periodontitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Dentaid SL (Industry)
Responsible Party: Principal Investigator, Dr. Melissa Fok, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P&ID2025-01
Record Dates: First submitted 2025-04-25; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Periodontitis; Periodontitis Stage II; Periodontitis Stage III
Keywords: Mouthwash; Chlorhexidine; CPC; Periodontitis; Mouthrinse; cetylpyridinium chloride; Oral antiseptic
MeSH Terms: conditions — Periodontitis | interventions — Chlorhexidine; Cetylpyridinium

STUDY DESIGN:
Intervention Model Description: randomized double blinded non-inferiority controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The allocation concealment will be maintained from all parties until data analysis stage.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active control (Active Comparator): CHX 0.2%
  Interventions: Other: Control (chlorhexidine with cetylpyridinium chloride)
- Experimental (Experimental): CHX 0.12%+CPC 0.05%
  Interventions: Other: Experimental (chlorhexidine)

INTERVENTIONS:
Other: Experimental (chlorhexidine) — Test group: administration of experimental antiseptic (CHX 0.12%+CPC 0.05%) for 3 weeks
  Arms: Experimental
Other: Control (chlorhexidine with cetylpyridinium chloride) — Active comparator: administration of control antiseptic (CHX 0.2%) for 3 weeks
  Arms: Active control

SUMMARY:
The focus of this study is on two types of mouthwashes - one containing a chlorhexidine (CHX) at 0.2% (CHX), and the other one containing CHX at a lower concentration of 0.12% with cetylpyridinium chloride (CPC). Both mouthwashes are used to help in the treatment of gum disease. CHX has been known for a long time for its effectiveness against plaque and mouth inflammation. It could inhibit and even kill them. However higher concentrations of CHX comes with unwanted side effect including altered taste, teeth staining and irritation in the mouth. Interestingly, these side effects seem to occur less frequently when a lower concentration CHX solution is used. CPC also combats bacteria by adhering quickly to the surfaces inside your mouth, although it has less substantivity than CHX, it has been shown to reduce plaque and gum inflammation effectively, and it typically causes fewer side effects than CHX. We hypothesize that this new formulation of CHX 0.12%+CPC mouthwash is non-inferior to CHX 0.2% in terms of its anti-plaque and anti-inflammatory properties while presenting with less side effects after 21 days of use. Microbiological samples and fluids from periodontal pockets will be collected before and after treatment for analysis of microbiological effects.

DETAILED DESCRIPTION:
* Aim: To compare the effects of 2 formulations of antiseptics on clinical efficacy (reduction of gingival inflammation and plaque) and oral microbiome when used as an adjuvant in periodontal treatment.
* Hypothesis: HA: The study mouthwash (CLX 0.12% + CPC 0.05%) when used as an adjunct to step 1 periodontal therapy, is non-inferior to control mouthwash (CHX 0.2%) in terms of inflammation and plaque control.
* Primary outcome: Changes in full mouth Bleeding on Probing (BoP) at 2 months after 21 days daily use of test mouthwash as an adjunct to step 1 periodontal therapy compared to active control.
* Secondary outcome:

Changes in BoP at 21 days after baseline. Changes in Löe and Silness Gingival Index at 21 days and 2 months after baseline.

Changes in modified O'Leary plaque index and Turesky modification of Quigley-Hein plaque index at 21 days, 2 months after baseline.

Changes in Tongue Coating Index and Lobene Stain Index at 14, 21 days and 2 months after baseline.

Pocket probing depth (PPD) and clinical attachment level (CAL) changes 2 months after baseline.

Subgingival microbiological changes at 21 days and 2 months after baseline. Gingival cervical fluid volume and inflammatory biomarker profile changes at 21 days and 2 months.

Taste alteration and mucosal irritation at 14 days, 21 days and 2 months after baseline.

Changes in patient-reported outcome measures at 21 days and 2 months after baseline

ELIGIBILITY:
Inclusion Criteria:

* Consenting patients with at least 6 evaluable teeth in each quadrant, including minimum 1 molar and 1 premolar.
* Generalized stage II-III periodontitis patients.
* Baseline BOP > 25%.
* No known allergy or adverse effects to CHX or CPC
* Non-smokers, non-orthodontic patients, no concurrent or past antibiotics/medication known to affect periodontal status (i.e. calcium antagonists, phenytoin)/anti-inflammatory therapy (i.e. NASIDs) in the last 3 months, pregnant/breastfeeding, compliance to study procedures.
* ASA class I-II patients.
* Either non-diabetic or with controlled diabetes (HbA1C<7).
* Normal/Elevated blood pressure (AHA - Systolic <130mmHg; Diastolic <80mmHg).
* No radiation/chemotherapy in the past 5 years
* No immunosuppression including drug induced immunosuppression.
* No participation in other clinical studies in the last 4 weeks.
* No administration of CHX or CPC in the last 3 months
* No periodontal treatment in the last 3 months.

Exclusion Criteria:

* Unable to provide written consent.
* Non-compliant study procedures.
* Patients with medical (including psychiatric) and pharmacotherapeutic histories that, in the investigator's opinion, may compromise the protocol.
* Patients requiring antibiotics prophylaxis for dental procedures.
* Patients with self-reported pregnancy or patients who are breastfeeding.
* Patients with history of use of systemic antibiotics, in combination with any form of periodontal treatment, within the past 3 months.
* Patients with uncontrolled endocrine disease.
* Patients who are not compliant with the review protocol, leading to deviation of more than 1 week.
* Patients requiring the admission of systemic antibiotics, in combination with any form of dental treatment, during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
% Bleeding on probing (BoP) | 2 months
  % BoP will be assessed at 6 surfaces (mesiobuccal, mid buccal, disto-buccal, mesio-oral, mid-oral, disto-oral.) in a dichotomous manner (Mühlemann & Son, 1971). Bleeding will be positive after 15 seconds of probing the gingival sulcus to the most apical stop. The percentage of the full mouth BoP will be reported.

SECONDARY OUTCOMES:
% Bleeding on probing (BoP) | 21 days
  % BoP will be assessed at 6 surfaces (mesiobuccal, mid buccal, disto-buccal, mesio-oral, mid-oral, disto-oral.) in a dichotomous manner (Mühlemann & Son, 1971). Bleeding will be positive after 15 seconds of probing the gingival sulcus to the most apical stop. The percentage of the full mouth BoP will be reported.
Macpherson modification of the Lobene Stain Index (MLSI) | 21 days and 2 months
  Tooth staining assessment by the Macpherson modification of the Lobene Stain Index (MLSI) (L. M. Macpherson, K. W. Stephen, A. Joiner, F. Schäfer, & E. Huntington, 2000) on index tooth (11, 12, 21, 22, 31, 32, 41, 42). If an incisor is missing, the nearest canine will serve as substitute where appropriate.
Full mouth plaque score | 21 days and 2 months
  Full Mouth Plaque Score (FMPS) (O'Leary et al., 1972) will be measured as an indicator of oral hygiene on the mesial, distal, buccal and oral surfaces of each tooth.
  The FMPS will be assessed with the following formula: Number of surfaces with plaque/Total number of surfaces x 100%
Clinical attachment level | 2 months
  CAL measures the distance from the cemento-enamel junction of the tooth to the base of the periodontal pocket.
  CAL will be measured at baseline and 2 months by recording the distance from the cervical line to the bottom of the probable pocket at 6 sites (Mesio-buccal, mid-buccal, disto-buccal, mesio-oral, mid-oral and disto-oral) for each of the study teeth.
Pocket probing depth (PPD) | 2 months
  PPD measures the distance from the free gingival margin to the base of the periodontal pocket. It will be measured at 6 sites (Mesio-buccal, mid-buccal, disto-buccal, mesio-oral, mid-oral and disto-oral) in the entire dentition.
Patient-reported outcome measures for mouthwash (PROMs-MW) | 14 days, 21 days, 2 months
  A mouthwash-specific questionnaire consisting of 6 questions was constructed to assess the compliance and potential side effects associated with mouthwash use, including burning sensation, altered taste and unpleasant taste assessed on a visual analogue scale., taking reference from Navabi and coworkers (Navabi, Afshari, Kamyabi, & Mohammadi, 2024). A higher score indicates a poorer patient-perceived experience.
Oral health impact profile for chronic periodontitis (OHIP-CP) | 21 days and 2 months
  Oral health impact profile for chronic periodontitis (OHIP-CP). The OHIP-CP is a condition-specific OHRQoL instrument for patients with chronic periodontitis consisting of 18 questions (He, Wang, Wei, & Ji, 2017). Fifteen questions from the OHIP-CP Cantonese version was adopted from the translated and validated Chinese version of OHIP (Wong, Lo, & McMillan, 2002). The remaining 3 questions were translated through forward translation, backward translation, expert committee process to reach a consensus. A higher score indicated poor oral health-related quality of life.
Löe and Silness Gingival Index | 21 days and 2 months
  Löe and Silness Gingival Index (1963) (Loe & Silness, 1963) will be performed on 4 gingival surfaces of index Ramfjord teeth (16, 21, 24, 36, 41, 44). Each of the four gingival areas (buccal, oral, mesial, distal) of the tooth is given a score from 0 to 3.
  The scores of the 4 areas will be added and divided by 4 to give the GI for the tooth The scores for individual teeth may be grouped to have the GI for the group of teeth Finally, by adding the indices for the teeth and dividing by the total number of teeth examined, the Gl for the individual is obtained. The index for the subject is thus an average score for the areas examined.
  Missing teeth from the Ramfjord index teeth (16, 21, 24, 36, 41, 44) will not be substituted.
Turesky modification of Quigley-Hein plaque index (TQHPI) | 21 days and 2 months
  Turesky modification of Quigley-Hein plaque index (TQHPI)(Turesky et al.,1970) on Ramfjord teeth (16, 21, 24, 36, 41, 44) will be performed.
  Each tooth will be divided into 6 surfaces (mesiobuccal, mid buccal, disto-buccal, mesio-oral, mid-oral, disto-oral.) Each surface will be given a score. The score of all sites will be summed and divided by the number of sites to have the individual tooth index The subject mean plaque score will be calculated by summing all the plaque indices of teeth and dividing by the number of teeth.
  Missing teeth from the Ramfjord index teeth (16, 21, 24, 36, 41, 44) will not be substituted.
Shannon or Simpson Diversity Index | 2 months
  This measure will assess the change in diversity of the microbial community in the sample (alpha diversity). A diversity index provides a mathematical measure that reflects the number of different species (richness) and the evenness of the species' abundances. It ranges from zero to infinity. A higher value means higer diversity.
Bray-Curtis Dissimilarity | 2 months
  It is a distance metrics that measures the beta-diversity. It quantifies the dissimilarity between microbial communitie/ the variation or differences in microbial communities between different samples. It ranges from 0 (identical communities) to 1 (completely different communities).
Biomarker concentrations from gingival cervicular fluid | 2 months
  The concentrations of a panel of biomarkers (IL-1β, TNF-α, IL-6, MMP-8,TIMP-1, TIMP-2) found within the gingival cervicular fluid (GCF) will be assessed with multiplex immunoassays. Unit: ng/mL or as appropriate based on assay's standard.

IPD SHARING:
Plan to Share IPD: No
There is concern that individual participant data sharing may violate data ownership policy of the institute. Information sheet and consent form approved by local IRB did not explicitly permit data sharing beyond the scope of the current study. As such, sharing IPD could potentially infringe upon the rights and expectations of our participants, which we are committed to safeguarding.